CLINICAL TRIAL: NCT05724550
Title: Diaphragm and Lung Ultrasound After Reversal of Rocuronium-induced Neuromuscular Blockade With Sugammadex or Neostigmine in Children Undergoing Surgery : A Randomized Double-blind Controlled Trial
Brief Title: Diaphragm Function After Reversal of Rocuronium-induced Neuromuscular Blockade With Sugammadex or Neostigmine in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ji-Hyun Lee, Clinical Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H2212-027-1383
Record Dates: First submitted 2023-01-15; First posted 2023-02-13 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Neuromuscular Block, Residual
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neostigmine (Active Comparator): The use of neostigmine 0.02mg/kg for reversal of neuromuscular blocking agent.
  Interventions: Drug: Neostigmine
- Sugammadex (Experimental): The use of sugammadex 2mg/kg for reversal of neuromuscular blocking agent.
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — * Sugammadex(100mg/mL), 2mg/kg
  * After confirming Train-of-four counts 4, patients allocated to sugammadex group receive sugammadex 2mg/kg for reversal of rocuronium at the end of the surgery.
  Other Names: bridion
  Arms: Sugammadex
Drug: Neostigmine — * Neostigmine methylsulfate(0.5mg/mL) 0.02mg/kg
  * After confirming Train-of-four counts 4, patients allocated to neostigmine group receive neostigmine 0.02mg/kg (maximum 5mg) combined with atropine 0.02mg/kg for reversal of rocuronium at the end of the surgery.
  Other Names: Neostigmine methylsulfate
  Arms: Neostigmine

SUMMARY:
This study is to evaluate the recovery of diaphragm function and atelectasis after reversal of neuromuscular blockade with Neostigmine and Sugammadex using lung ultrasound and diaphragm ultrasound for children aged 2 to 7 who are scheduled for the surgical procedure under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 2 and 7 who are scheduled for surgery lasting more than 1 hour under general anesthesia using a neuromuscular blocking agent

Exclusion Criteria:

* Patients with a history of severe respiratory disease with a high risk of bronchoconstriction
* Patients with abnormal findings on preoperative chest radiography such as severe atelectasis, pneumothorax, pleural effusion, or pneumonia.
* Patients with severe renal or liver disease, or neuromuscular disease
* Patients with a history of allergy to drugs (sugammadex, rocuronium neostigmine)
* Patients with significant bradycardia
* Patients scheduled for surgery where estimated blood loss during surgery is expected to be more than 30% of estimated blood volume, or cases where fluid imbalance is expected to be severe during surgery
* patients scheduled for lung parenchyme/diaphragm/thoracic surgery
* other researchers considered it inappropriate to participate in research.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-08 (Actual)

PRIMARY OUTCOMES:
Diaphragm excursion ratio | during diaphragm ultrasound procedure after reversal of neuromuscular blocking agent (T1), an average of 10 minute
  The ratio of diaphragm excursion at the time before injecting neuromuscular blocking agent before surgery (T0) and diaphragm excursion at the time after reversal of neuromuscular blocking agent (T1)

SECONDARY OUTCOMES:
modified lung ultrasound score before neuromuscular blockade (LUS_T0) | during lung ultrasound procedure before neuromuscular blocking agent (T0), an average of 10 minutes
  Both lung ultrasound score can be calculated by adding up the 12 individual pulmonary quadrant scores yielding a score between 0 (no aeration loss) and 36 (complete aeration loss)
modified lung ultrasound score after reversing neuromuscular blockade (LUS_T1) | during lung ultrasound procedure after reversing neuromuscular blocking agent(T1), an average of 10 minutes
  Both lung ultrasound score can be calculated by adding up the 12 individual pulmonary quadrant scores yielding a score between 0 (no aeration loss) and 36 (complete aeration loss)
modified lung ultrasound score at post-anesthesia care unit (PACU) (LUS_T2) | 30 minutes after entering the post-anesthesia care unit (T2)
  Both lung ultrasound score can be calculated by adding up the 12 individual pulmonary quadrant scores yielding a score between 0 (no aeration loss) and 36 (complete aeration loss)
total recovery time (sec) | From injection of neuromuscular block reversal agent to extubation, not to exceed 20 minutes
  time from injection of a neuromuscular block reversal agent to extubation
perioperative respiratory adverse events | intraoperative
  laryngospasm, bronchospasm, desaturation (SpO2 < 95%), airway obstruction, severe coughing, postoperative stridor during the emergence period
length of stay in post-anesthesia care unit | from entering the post-anesthesia care unit to discharge from the post-anesthesia care unit, up to 24 hours
  Length of stay in post-anesthesia care unit
Adverse events occurred during post-anesthesia care unit stay | from entering the post-anesthesia care unit to discharge from the post-anesthesia care unit, up to 24 hours
  agitation, stridor, desaturation (SpO2<95%), nausea, vomiting, bradycardia, somnolence, need for oxygen support
postoperative pulmonary complication | from entering the general ward after surgery to discharge from hospital, up to 7 days
  pneumonia, respiratory failure, pleural effusion, atelectasis described in postoperative chest radiography, pneumothorax, bronchospasm, aspiration pneumonia

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongrogu, South Korea

REFERENCES:
- [Derived] Park JB, Kim TW, Ji SH, Jang YE, Kim EH, Kim JT, Kim HS, Lee JH. Ultrasonographic assessment of sugammadex-enhanced early recovery of diaphragmatic function in children: A randomised double-blind controlled trial. Eur J Anaesthesiol. 2025 Oct 1;42(10):907-915. doi: 10.1097/EJA.0000000000002231. Epub 2025 Jul 7. PMID 40625141